CLINICAL TRIAL: NCT00814086
Title: A Phase I Feasibility Trial IP Cisplatin and IV Paclitaxel on Day 1 Followed by IP Paclitaxel on Day 8 Every 21 Days as Front-Line Treatment of Ovarian, Fallopian Tube and Primary Peritoneal Carcinoma
Brief Title: Cisplatin and Paclitaxel in Treating Patients With Stage IIB, Stage IIC, Stage III, or Stage IV Ovarian Epithelial Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cavity Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-9921; NCI-2009-00624 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG-9921; CDR0000629746; GOG-9921 (Other: Gynecologic Oncology Group); GOG-9921 (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2008-12-20; First posted 2008-12-23 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Chemotherapeutic Agent Toxicity; Endometrial Adenocarcinoma; Fallopian Tube Carcinoma; Gastrointestinal Complication; Malignant Ovarian Mixed Epithelial Tumor; Neurotoxicity Syndrome; Ovarian Brenner Tumor; Ovarian Clear Cell Cystadenocarcinoma; Ovarian Mucinous Cystadenocarcinoma; Ovarian Serous Cystadenocarcinoma; Primary Peritoneal Carcinoma; Stage II Ovarian Cancer; Stage III Ovarian Cancer; Stage IV Ovarian Cancer; Undifferentiated Ovarian Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Neurotoxicity Syndromes; Brenner Tumor; Ovarian Neoplasms | interventions — Paclitaxel; Taxes; Cisplatin

ARMS (1):
- Treatment (paclitaxel, cisplatin) (Experimental): Patients receive paclitaxel IV over 3 hours and cisplatin intraperitoneally (IP) on day 1 and paclitaxel IP on day 8. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Paclitaxel; Drug: Cisplatin

INTERVENTIONS:
Drug: Paclitaxel — Given IV or intraperitoneally
  Other Names: Anzatax; TAX
Drug: Cisplatin — Given intraperitoneally

SUMMARY:
This phase I trial is studying the side effects and best dose of cisplatin given together with paclitaxel in treating patients with stage IIB, stage IIC, stage III, or stage IV ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cavity cancer. Drugs used in chemotherapy, such as cisplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) and giving them in different ways may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the feasibility of intraperitoneal (IP) cisplatin and intravenous (IV) paclitaxel followed by IP paclitaxel in patients with stage IIB, IIC, III, or IV ovarian epithelial, fallopian tube, or primary peritoneal cavity cancer.

SECONDARY OBJECTIVES:

I. Assess the toxicity of this regimen in these patients. II. Determine the types of surgical and catheter complications that may occur after surgery or during the course of treatment in these patients.

III. Estimate the response rate in patients with measurable disease treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive paclitaxel IV over 3 hours and cisplatin intraperitoneally (IP) on day 1 and paclitaxel IP on day 8. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed ovarian epithelial, fallopian tube, or primary peritoneal cavity cancer

  * Stage IIB, IIC, III, or IV disease
  * Optimal or suboptimal residual disease after debulking surgery within the past 12 weeks

    * Appropriate tissue for histologic evaluation available
* The following histologic epithelial cell types are eligible:

  * Serous adenocarcinoma
  * Endometrioid adenocarcinoma
  * Mucinous adenocarcinoma
  * Undifferentiated carcinoma
  * Clear cell adenocarcinoma
  * Mixed epithelial carcinoma
  * Transitional cell carcinoma
  * Malignant Brenner tumor
  * Adenocarcinoma not otherwise specified
  * Carcinosarcoma
* No ovarian epithelial carcinoma of low malignant potential (borderline carcinomas)
* No synchronous primary endometrial cancer or a history of primary endometrial cancer unless all of the following conditions are met:

  * Stage ≤ IB disease
  * No more than superficial myometrial invasion, without vascular or lymphatic invasion
  * No poorly differentiated subtypes, including papillary serous, clear cell, or other FIGO grade 3 lesion
* GOG performance status 0-2
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Serum creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* SGOT ≤ 2.5 times ULN
* Audiograms required after study chemotherapy courses 3 and 6 for patients with hearing loss, or who are experiencing tinnitus during study therapy
* Negative pregnancy test
* Not pregnant or nursing
* Fertile patients must use effective contraception
* None of the following:

  * Septicemia
  * Severe infection requiring parenteral antibiotics
  * Malnutrition requiring parenteral hyperalimentation
  * Acute hepatitis
  * Any other major medical conditions expected to interfere with completion of protocol therapy
* No active bleeding
* No circumstances that would prohibit completion of study therapy or required follow-up
* No history of allergic reaction to polysorbate 80 (e.g., etoposide or vitamin E)
* No other invasive malignancies, except for nonmelanoma skin cancer or other specific malignancies within the past 5 years, or whose previous cancer treatment contraindicates this protocol therapy
* No unstable angina or myocardial infarction within the past 6 months

  * Abnormal cardiac conduction (e.g., bundle branch block or heart block) that has been stable for the past 6 months allowed
* No prior targeted therapy for the management of ovarian epithelial or primary peritoneal cavity cancer including, but not limited to, the following:

  * Vaccines
  * Antibodies
  * Tyrosine kinase inhibitors
* No prior chemotherapy
* No prior radiotherapy
* No prior hormonal therapy for the management of epithelial ovarian or primary peritoneal cavity cancer

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-02; Primary Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Number of patients who have at least 1 dose-limiting toxicity or delay in therapy for more than 2 weeks | 12 weeks

SECONDARY OUTCOMES:
Grade of toxicity as assessed by Common Terminology Criteria for Adverse Events version 3.0 (CTCAE v3.0) | Up to 1 year
Adverse events related to the catheter or the surgical placement of the catheter | Up to 1 year
Objective tumor response (partial or complete) assessed by Response Evaluation Criteria for Solid Tumors (RECIST) | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Don Dizon, Principal Investigator — Gynecologic Oncology Group
Locations (7):
- United States (7):
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Riverside Methodist Hospital, Columbus, Ohio
  - Tulsa Cancer Institute, Tulsa, Oklahoma
  - Women and Infants Hospital, Providence, Rhode Island
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin